CLINICAL TRIAL: NCT00736814
Title: Genotype-driven Treatment of Advanced Non-small Cell Lung Cancer Based on mRNA Expression of ERCC1 & RRM1 as First-line Chemotherapy
Brief Title: First-Line Combination Chemotherapy in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer That Cannot Be Removed by Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000609880; YONSEI-4-2008-0132; SANOFI-AVENTIS-YONSEI-4-2008-0
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2009-08

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Docetaxel; Gemcitabine; Vinorelbine

ARMS (5):
- Arm I (Active Comparator): Patients receive standard chemotherapy of docetaxel and carboplatin.
  Interventions: Drug: carboplatin; Drug: docetaxel
- Arm II, Genotype A1 (Experimental): Patients receive docetaxel and vinorelbine ditartrate.
  Interventions: Drug: docetaxel; Drug: vinorelbine tartrate
- Arm II, Genotype A2 (Experimental): Patients receive gemcitabine hydrochloride and vinorelbine ditartrate.
  Interventions: Drug: gemcitabine hydrochloride; Drug: vinorelbine tartrate
- Arm II, Genotype B1 (Experimental): Patients receive docetaxel and carboplatin.
  Interventions: Drug: carboplatin; Drug: docetaxel
- Arm II, Genotype B2 (Experimental): Patients receive gemcitabine hydrochloride and carboplatin.
  Interventions: Drug: carboplatin; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: carboplatin — Given intravenously
  Arms: Arm I; Arm II, Genotype B1; Arm II, Genotype B2
Drug: docetaxel — Given intravenously
  Arms: Arm I; Arm II, Genotype A1; Arm II, Genotype B1
Drug: gemcitabine hydrochloride — Given intravenously
  Arms: Arm II, Genotype A2; Arm II, Genotype B2
Drug: vinorelbine tartrate — Given intravenously
  Arms: Arm II, Genotype A1; Arm II, Genotype A2

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known which combination chemotherapy regimen is most effective in treating non-small cell lung cancer.

PURPOSE: This randomized phase II trial is comparing different combination chemotherapy regimens to see how well they work as first-line therapy in treating patients with stage IIIB or stage IV non-small cell lung cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess treatment outcomes of adjuvant chemotherapy based on ERCC1 and RRM1 mRNA levels in patients with stage IIIB or IV non-small cell lung cancer.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

RNA is isolated from pretreatment biopsy samples and analyzed with reverse transcriptase-PCR (RT-PCR) assays to determine ERCC1 and RRM1 mRNA expression.

* Arm I: Patients receive standard chemotherapy comprising docetaxel IV and carboplatin IV on day 1. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients are treated according to ERCC1 and RRM1 mRNA expression levels as determined by RT-PCR.

  * Genotype A1 (high ERCC1 and high RRM1 mRNA levels): Patients receive non-platinum doublet chemotherapy comprising docetaxel and vinorelbine ditartrate IV on days 1 and 15. Treatment repeats every 4 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  * Genotype A2 (high ERCC1 and low RRM1 mRNA levels): Patients receive non-platinum doublet chemotherapy comprising gemcitabine hydrochloride IV and vinorelbine ditartrate IV on days 1 and 8. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  * Genotype B1 (low ERCC1 and high RRM1 mRNA levels): Patients receive platinum doublet chemotherapy comprising docetaxel IV and carboplatin IV on day 1. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  * Genotype B2 (low ERCC1 and low RRM1 mRNA levels): Patients receive platinum doublet chemotherapy comprising gemcitabine hydrochloride IV on days 1 and 8 and carboplatin IV on day 1. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven or radiologically and clinically suspected stage IIIB (with malignant pleural effusion) or IV non-small cell lung cancer
* Unresectable disease
* At least 1 measurable lesion (> 10 mm with spiral CT scan or > 20 mm with conventional CT scan)
* No symptomatic or untreated brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 12 weeks
* ANC ≥ 1,500/mm³
* Hemoglobin > 9.0 g/dL
* Platelet count ≥ 100,000/mm³
* AST and ALT < 2 times upper limit of normal (ULN)
* Bilirubin < 1.5 mg/dL
* Creatinine < 1.5 times ULN
* Not pregnant or nursing
* No serious uncontrolled systemic intercurrent illness, including any of the following:

  * Acute myocardial infarction
  * Uncontrolled arrhythmia
  * Uncontrolled heart failure
  * Sepsis
  * Poorly controlled diabetes
* No other malignancy within the last 5 years, except for carcinoma in situ of the cervix or nonmelanomatous carcinoma of the skin

PRIOR CONCURRENT THERAPY:

* At least 3 weeks since prior radiotherapy, including cranial irradiation
* At least 3 weeks since prior major surgery
* No prior systemic chemotherapy except adjuvant chemotherapy provided it was completed more than 12 months ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2008-06

PRIMARY OUTCOMES:
Response rate (complete and partial responses)

SECONDARY OUTCOMES:
Disease control rate
Response duration
Progression-free survival
Overall survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Byung Chul Cho, Principal Investigator — Yonsei University
Locations (1):
- Yonsei Cancer Center at Yonsei University Medical Center, Seoul, South Korea